# Statistical Design and Power

ClinicalTrials.gov Identifier: NCT05187013

Unique Protocol ID: NCR203140

Title: mHealth to Address Uncontrolled Hypertension Among Hypertensive Homeless Adults

Version Date: January 26, 2021

### STATISTICAL DESIGN AND POWER

## Sample size and statistical power:

The study is powered for the outcomes of AIM 2 and based on the comparison of mean BP between the CL and INT groups at 6 months. Given the data scarcity on the effect of mHealth strategy on HTN in the PEH, there is not sufficient data for power estimation. A decrease in SBP of 5 mmHg is associated with clinically important reduction in the relative risk of stroke/CAD events (66). Based on our recent study (14), we used the standard deviation of SBP (15 mmHg) and DBP (13 mmHg) to calculate sample size. Assuming a two-sample *t*-test, we calculated that a total of 120 (60 per each group) is sufficient to achieve a power of 80% to detect a difference of 8 mmHg assuming the SD for both groups is at 15 at the 0.05 significance level (two-sided). Based on data from our site, this is a conservative power estimate for either outcome of SBP or DBP. Up to 27% of PEH have HTN (6); 40% uncontrolled (14). In 2019, the PR served at least 1000 unique PEH with HTN (53). Using medical record reviews and outreach, with a conservative 50% response rate, we will be able to enroll 120 participants within 4-6 months. Risk of contamination will be low as weekly enrollment in each clinic is low and PEH are from different shelters (each 100-300 PEH) in and outside PR or on streets.

# **Data Analysis, Outcomes and Measurements:**

<u>AIM 1</u>: The primary outcomes are changes in SBP and DBP and the percentage/degree of adherence to BP medications and appointment attendance.

Blood pressure will be measured by clinic nurses at the initial enrollment and at each follow ups to the end of study follow-up period for each participant. BPs will be measured with the patient seated in an upright position with right arm resting on a table at the level of heart and a proper cuff size is fitted, after 5 min rest (60). Since patients are already diagnosed with HTN, BP readings from the most recent visit will be used to determine uncontrolled vs controlled HTN. Uncontrolled BP is defined based on the current updated guideline (SBP>140 or DPB>90 mmHg) and considering other co-morbidity including CAD, stroke, MI, DM or chronic kidney disease (54). When no co-morbidity, we define Stage 2/Uncontrolled HTN as ≥140/90<160/100, and "Stage 3/Very uncontrolled ≥160/100".

Adherence to medication for each participant will be measured by Voils DOSE-nonadherence tool (68,69). Appointment attendance is collected via medical records and as ratio and number of kept appointments to all appointments scheduled (0-100%) (58). Other outcomes will include utilization and frequency of phone and SMS text use/message exchanges for the level of engagement (number of texts read and responded by participants) (58); phone retention rates; changes in adherence to other CVD medications (statin, anti-platelets) and risk factors (non-HDL or LDL, smoking cessation); (56,57). Interim analysis will be performed. Final analysis will be performed after the completion of data collection. Main predictor is the HTN specific mHealth intervention. Independent variables including self-reported sociodemographic and clinical data/indicators (including age, race/ethnicity, gender, years and episodes of homelessness, BMI, health insurance status, and history of chronic disease such as diabetes, renal insufficiency, hyperlipidemia, asthma, COPD and CAD/MI, tobacco, alcohol or substance abuse, or mental illness), will be analyzed for the association with the outcomes.

<u>AIM 2</u>: Attitudes, acceptance and experience of mHealth will be assessed from qualitative individual audiotaped interviews with hypertensive patients and providers using 8-10 open-ended questions with probes. Primary discussions with key informants in the shelters for discourse will help bring up issues to be explored by questions during interviews.

## **Analytic Plan and Statistical Analysis:**

**AIM 1:** The primary statistical analysis will be on an intention-to-treat basis. The trial results will be reported as comparative summary statistics (difference in response rate or means) with 95% confidence intervals and in accordance with the CONSORT. All statistical tests will use a 0.05 two-sided significance level. We will test the difference of outcomes (change in SBP and DBP from baseline) between the groups after 6 months using a two-sample t-test. We will examine the outcomes using a mixed-effects model on data collected at 6 months to calculate the outcome of change from baseline. An interaction between time and randomized group will be fitted

to allow estimation of treatment effects (INT vs. CL) at each time point. Analysis of covariance will be used in place of a t-test, if covariates needed. A regression analysis will be performed using the final assessment of adherence as a response and randomization group as a predictor. Other variables that may potentially have effects on adherence such as age, gender, education and comorbidity will also be included if they are not balanced between groups by the randomization or if determined by univariate analysis to be significantly predictive of adherence. The medication adherence will be calculated for 6 months and compared between two groups using the generalized estimation equation (GEE) method (or multivariate ANOVA). Message exchanges in two groups will be analyzed for the engagement level to explain outcomes. Numbers and percentages of appointment attendance and all secondary outcomes will be compared between groups. We will report missing data and explore patterns and mechanism, though a mixed-effects model does implicitly account for data missing at random. We will report all results in total numbers and percentages.

**AIM 2:** Interviews will be transcribed coded and analyzed using an inductive grounded theory analysis. Content analysis will be done by two research team members to identify core perceptions regarding mHealth strategy for HTN management. During content analysis, we will develop preliminary coding based on priority codes derived from the theoretical framework and conceptual model guiding the study. We will perform critical deliberation about initial coding and review coding for similarities and variations among coders' output to achieve a high level of agreement and assure that the coding scheme is appropriate. Reviewers will independently review codes, meet and discuss them, identify concepts and categories, and describe major important themes.

### Reference:

- 1. National Alliance to End Homelessness. The State of Homelessness in America 2020. (accessed June 2, 2020). Available at https://endhomelessness.org/homelessness-in-america/homelessness-statistics/state-ofhomelessness-2020
- 2. National Alliance to End Homelessness. The State of Homelessness in America 2013. Homeless Research Institute. Accessed June 2 2020, available at http://www.ncdsv.org/images/NAEH\_StateOfHomelessnessInAmerica\_4-2013.pdf
- 3. Fargo J, Metraux S, Byrne T, Munley E, Montgomery AE, Jones H, Sheldon G, Kane V, Culhane D. Prevalence and Risk of Homelessness Among US Veterans. Prev Chronic Dis. 2012; 9: E45. Epub 2012 Jan 26.
- 4. Culhane DP, Metraux S, Byrne T, Stino M, Bainbridge J. The age structure of contemporary homelessness: evidence and implications for public policy. Analyses of Social Issues and Public Policy, 2013 Jan, DOI:10.1111/asap.12004. available at https://spssi.onlinelibrary.wiley.com/doi/abs/10.1111/asap.12004
- 5. Kushel MB, Vittinghoff E, Haas JS. "Factors associated with the health care utilization of homeless persons." JAMA. 2001 Jan 10;285(2):200-6.
- 6. Bernstein, R. S., Meurer, L. N., Plumb, E. J., & Jackson, J. L. Diabetes and hypertension prevalence in homeless adults in the United States: a systematic review and meta-analysis. Am J Public Health, 2015;105(2): e46-e60.
- 7. Gelberg L1, Linn LS. Assessing the physical health of homeless adults. JAMA. 1989 Oct 13;262(14):1973-9.
- 8. Szerlip MI1, Szerlip HM. dentification of cardiovascular risk factors in homeless adults. Am J Med Sci. 2002 Nov;324(5):243-6.
- 9. Moczygemba LR1, Kennedy AK, Marks SA, Goode JV, Matzke GR. A qualitative analysis of perceptions and barriers to therapeutic lifestyle changes among homeless hypertensive patients. Res Social Adm Pharm. 2013 Jul-Aug;9(4):467-81. doi: 10.1016/j.sapharm.2012.05.007. Epub 2012 Jul 25.
- Kim DH1, Daskalakis C, Plumb JD, Adams S, Brawer R, Orr N, Hawthorne K, Toto EC, Whellan DJ. Modifiable cardiovascular risk factors among individuals in low socioeconomic communities and homeless shelters. Fam Community Health. 2008 Oct-Dec;31(4):269-80. doi: 10.1097/01.FCH.0000336090.37280.2e.
- 11. Savage CL1, Lindsell CJ, Gillespie GL, Dempsey A, Lee RJ, Corbin A. Health care needs of homeless adults at a nurse-managed clinic. J Community Health Nurs. 2006 Winter;23(4):225-34.
- 12. Kleinman LC, Freeman H, Perlman J, Gelberg L. Homing in on the homeless: assessing the physical health of homeless adults in Los Angeles County using an original method to obtain physical examination data in a survey. Health Serv Res. 1996 Dec;31(5):533-49.
- 13. Lee TC1, Hanlon JG, Ben-David J, Booth GL, Cantor WJ, Connelly PW, Hwang SW. Risk factors for cardiovascular disease in homeless adults. Circulation. 2005 May 24;111(20):2629-35. Epub 2005 May 16.

- 14. Asgary R, Sckell B, Alcabes A, Naderi R, Schoenthaler A, Ogedegbe G. Rates and predictors of uncontrolled hypertension among hypertensive adults using New York City shelter-based clinics. Ann Fam Med. Jan-Feb 2016;14(1):41-6
- 15. Joffres M, Falaschetti E, Gillespie C, Robitallie C, Loustalot F, Poulter N, McAlister FA, Johansen H, Baclic O, Campbell N. Hypertension prevalence, awareness, treatment and control in national surveys from England, the USA and Canada, and correlation with stroke and ischemic heart disease mortality: a cross-sectional study. BMJ Open. 2013 Aug 30;3(8):e003423.doi:10.1136/bmjopen-2013003423.
- 16. Khandor E, Mason K, Chambers C, Rossiter K, Cowan L, Hwang SW. Access to primary health care among homeless adults in Toronto, Canada: results from the Street Health survey. *Open Med* 2011;5(2): e94e103.
- 17. Baggett TP1, Hwang SW, O'Connell JJ, Porneala BC, Stringfellow EJ, Orav EJ, Singer DE, Rigotti NA. Mortality among homeless adults in Boston: shifts in causes of death over a 15-year period. JAMA Intern Med. 2013 Feb 11;173(3):189-95. doi: 10.1001/jamainternmed.2013.1604.
- 18. Hwang SW, Orav EJ, O'Connell JJ, Lebow JM, Brennan TA. Causes of death in homeless adults in Boston. Ann Intern Med. 1997 Apr 15;126(8):625–628.
- 19. Appel LJ, Brands MW, Daniels SR, Karanja N, Elmer PJ, Sacks FM. Dietary approaches to prevent and treat hypertension: a scientific statement from the American Heart Association. *Hypertension*. Feb 2006;47(2):296-308.
- 20. Appel LJ, Champagne CM, Harsha DW, et al. Effects of comprehensive lifestyle modification on blood pressure control: main results of the PREMIER clinical trial. *JAMA*. Apr 23-30 2003;289(16):2083-2093.
- 21. Stamler R, Stamler J, Grimm R, et al. Nutritional therapy for high blood pressure. Final report of a four-year randomized controlled trial--the Hypertension Control Program. *JAMA*. Mar 20 1987;257(11):1484-1491.
- 22. Taylor E, Lake, T., Nysenbaum, J., Peterson, G., Meyers, D. Coordinating Care in the Medical Neighborhood: Critical Components and Available Mechanisms. Agency for Healthcare Research and Quality; 2011. AHRQ Publication No.11-0064. available at <a href="https://pcmh.ahrq.gov/page/coordinating-care-medicalneighborhood-critical-components-and-available-mechanisms">https://pcmh.ahrq.gov/page/coordinating-care-medicalneighborhood-critical-components-and-available-mechanisms</a>
- 23. Pham HH. Good neighbors: how will the patient-centered medical home relate to the rest of the health-care delivery system? *J Gen Intern Med.* Jun;25(6):630-634.
- 24. Gurol-Urganci I, de Jongh T, Vodopivec-Jamsek V, Atun R, Car J. Mobile phone messaging reminders for attendance at healthcare appointments. *Cochrane Database Syst Rev.* 2013, dec 5;2013(12): CD007458. DOI:
- 10.1002/14651858.CD007458.pub3. available at <a href="https://pubmed.ncbi.nlm.nih.gov/24310741/">https://pubmed.ncbi.nlm.nih.gov/24310741/</a>
- 25. Guy R, Hocking J, Wand H, Stott S, Ali H, Kaldor J. How effective are short message service reminders at increasing clinic attendance? A meta-analysis and systematic review. Health Serv Res. 2012 Apr;47(2):614-32.
- 26. Márquez Contreras E1, de la Figuera von Wichmann M, Gil Guillén V, Ylla-Catalá A, Figueras M, Balaña M, Naval J. Effectiveness of an intervention to provide information to patients with hypertension as short text messages and reminders sent to their mobile phone (HTA-Alert)]. Aten Primaria. 2004 Nov 15;34(8):399-405.

- 27. McGillicuddy JW, Gregoski MJ, Weiland AK, Rock RA, Brunner-Jackson BM, Patel SK, Thomas BS, Taber DJ, Chavin KD, Baliga PK, Treiber FA. Mobile Health Medication Adherence and Blood Pressure Control in Renal Transplant Recipients: A Proof-of-Concept Randomized Controlled Trial. JMIR Res Protoc. 2013 Sep 4;2(2):e32.
- 28. Hamine S, Gerth-Guyette E, Faulx D, Green BB, Ginsburg AS. Impact of mHealth chronic disease management on treatment adherence and patient outcomes: a systematic review. J Med Internet Res. 2015 Feb 24;17(2):e52. doi: 10.2196/jmir.3951.
- 29. Dick JJ, Nundy S, Solomon MC, Bishop KN, Chin MH, Peek ME. Feasibility and usability of a text message-based program for diabetes self-management in an urban African-American population. J Diabetes Sci Technol. 2011 Sep 1;5(5):1246-54.
- 30. DeKoekkoek T, Given B, Given CW, Ridenour K, Schueller M, Spoelstra SL.mHealth SMS text messaging interventions and to promote medication adherence: an integrative review. J Clin Nurs. 2015 Oct;24(1920):2722-35. doi: 10.1111/jocn.12918. Epub 2015 Jul 27.
- 31. Marcum ZA, Sevick MA, Handler S. Medication Nonadherence, A diagnosable and Treatable Medical Condition. JAMA, May 2013; 309 (20):2015-6
- 32. Viswanathan M, Golin CE, Jones CD, et al. Interventions to improve adherence to self-administered medications for chronic diseases in the United States: a systematic review. Ann Intern Med. 2012;157(11):785795.
- 33. Post LA, Vaca FE, Doran KM, Luco C, Naftilan M, Dziura J, Brandt C, Bernstein S, Jagminas L, D'Onofrio G. New media use by patients who are homeless: the potential of mHealth to build connectivity. J Med Internet Res. 2013 Sep 3;15(9):e195. doi: 10.2196/jmir.2724.
- 34. Eyrich-Garg KM. Mobile phone technology: a new paradigm for the prevention, treatment, and research of the non-sheltered "street" homeless? J Urban Health. 2010 May;87(3):365-80.
- 35. Asgary R, Sckell B, Alcabes A, Naderi R, Adongo P, Ogedegbe G. Perceptions, attitudes, and experience regarding mHealth among homeless. J Health Commun. 2015;20(12):1473-80
- 36. Jennings L, Lee N, Shore D, Strohminger N, Allison B, Conserve D, Cheskin LJ. US. Minority Homeelss Youth's Access to and Use of Mobile Phones: Implications for Health Intervention Design. J Health Commun. 2016;21(7):725-33
- 37. McInnes DK, Petrakis BA, Gifford AL, Rao SR, Houston TK, Asch STM, O'Toole TP. Retaining Homeless Veterans in Outpatient Care: A Pilot Study of Mobile Phone Text Message Appointment Reminders. AM J Public Health. 2014;104 suppl:s588-94.doi:10.2105/AJPH.2014.302061
- 38. Clover AC, Schueller SM, Winiarski DA, Smith DL, Karnik NS, Zalta A. Automated Mobile Phone-Based Mental Health Resource for Homeelss Youth: Pilot Study Assessing Feasibility and Acceptability. JMIR Ment Health. 2019;6(10):e1511.doi:10.2196/15144
- 39. Foyabo J, Bessetti-Barrett C. Improving clinic attendance through text message reminders to homeless patients with chronic health conditions. 2019, accessed June 2, 2020, available at <a href="https://www.elitecme.com/resource-center/health-information-professionals/improving-clinic-attendancethrough-text-message-reminders-to-homeless-patients-with-chronic-health-conditions/">https://www.elitecme.com/resource-center/health-information-professionals/improving-clinic-attendancethrough-text-message-reminders-to-homeless-patients-with-chronic-health-conditions/</a>
- 40. Prochaska, J. O. & Prochaska, J. M. Helping cure health care systems: Changing minds and behaviour.

Disease Management and Health Outcomes, Medicine, Published 1999, *6*, 335-341, DOI.10.2165/00115677199906060-0004

- 41. Johnson SS, Driskell MM, Johnson JL, Prochaska JM, Zwick W, Prochaska JO. Efficacy of a transtheoretical model-based expert system for antihypertensive adherence. Dis Manag. 2006 Oct;9(5):291301.
- 42. Glasgow RE, Orleans CT, Wagner EH. Does the chronic care model serve also as a template for improving prevention? *Milbank Quarterly.* 2001;79(4):579-612, iv-v.
- 43. Tsai AC, Morton SC, Mangione CM, Keeler EB. A meta-analysis of interventions to improve care for chronic illnesses. *Am J Manag Care*. Aug 2005;11(8):478-488.
- 44. Wagner EH. Chronic disease management: what will it take to improve care for chronic illness? Eff Clin Pract. 1998;1:2-4
- 45. Asgary R, Garland V, Jakubowski A, Sckell B. Colorectal cancer screening among the homeless population of New York City shelter-based clinics. Am J Pub Health. 2014;104(7):1307-13
- 46. Chen ZW, Fang LZ, Chen LY, Dai HL. Comparison of an SMS text messaging and phone reminder to improve attendance at a health promotion center: a randomized controlled trial. J Zhejiang Univ Sci B. 2008 Jan;9(1):34-8.
- 47. Leong KC, Chen WS, Leong KW, Mastura I, Mimi O, Sheikh MA, Zailinawati AH, Ng CJ, Phua KL, Teng CL. The use of text messaging to improve attendance in primary care: a randomized controlled trial. Fam Pract. 2006 Dec;23(6):699-705.
- 48. National Health Care for the Homeless Council. Training and Technical Assistance. Telehealth Webinars, Using Telehealth to manage Diabetes (2020), Tele-Behavioral Health in Homeless Health Care; Why Is it Hard, and What Can we DO About it? (2019), Accessed June 2<sup>nd</sup> 2020, available at <a href="https://nhchc.org/clinical-practice/homeless-services/telehealth/">https://nhchc.org/clinical-practice/homeless-services/telehealth/</a>
- 49. Iheanacho T, Payne K, Tsai J. Mobile, Community-Based buprenorphine Treatment for Veterans Experiencing Homelessness With Opioid Use Disorder: A Pilot, Feasibility Study. Am J Addict. 2020;doi.10.1111/ajad.13055.Online ahead of print
- 50. Gong K, Yan YL, Li Y, Du J, Wang J, Han Y, Zou Y, Z XY, Huang H, She Q. Mobile Health Applications for the Management of Primary Hypertension: A multicenter, Randomized, Controlled Trial. *Medicine*. 2020;99(16):e19715
- 51. How many people experience homelessness? NCH Fact Sheet No. 2. National Coalition for the Homeless Web site. February 2013. (accessed June 2, 2020) http://www.nationalhomeless.org/factsheets/How Many.pdf
- 52. The 2011 Annual Homeless Assessment Report to Congress. Nov 2012. The US Department of Housing and Urban Development Office of Community Planning and Development. (accessed June 2, 2020) <a href="https://www.onecpd.info/resources/documents/2011AHAR FinalReport.pdf">https://www.onecpd.info/resources/documents/2011AHAR FinalReport.pdf</a>
- 53. Project Renewal. What We Do. Accessed June 2, 2020, available at <a href="https://www.projectrenewal.org/programs-overview">https://www.projectrenewal.org/programs-overview</a>
- 54. Whelton PK, Carey RM, Aronow WS et al. 2017

ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice. J Am Coll Cardiol. 2018;71(19):2199-2269. Available at

https://www.onlinejacc.org/content/71/19/2199? ga=2.76732177.505114254.15922621811057634203.1592262181

- 55. Bobrow K, Brennan T, Springer D, Levitt NS, Rayner B, Namane M, Yu LM, Tarassenko L, Farmer A. Efficacy of a text messaging (SMS) based intervention for adults with hypertension: protocol for the StAR (SMS Text-message Adherence suppoRt trial) randomised controlled trial. *BMC Public Health*. 2014 Jan 11;14:28. doi: 10.1186/1471-2458-14-28.
- 56. Million Hearts. Tools & Protocols. Accessed June 2, 2020, available at https://millionhearts.hhs.gov/toolsprotocols/index.html
- 57. Richards AK, Jackson NJ, Cheng EM, Bryg RJ, Brown A, Towfighi A, Sanossian N, Barry F, Li N.

Derivation and Application of a Tool to Estimate Benefits From Multiple Therapies That Reduce Recurrent Stroke Risk. *Stroke*.2020;51(5):1563-1569

- 58. McInnes DK. Self- management Using text Messaging in a Homeless Population. ClinicalTrial.gov. Accessed June 2, 2020, available at https://clinicaltrials.gov/ct2/show/record/NCT03034993
- 59. Guy R, Hocking J, Wand H, Stott S, Ali H, Kaldor J. How effective are short message service reminders at increasing clinic attendance? A meta-analysis and systematic review. Health Serv Res. 2012 Apr;47(2):614-32.
- doi: 10.1111/j.1475-6773.2011.01342.x
- 60. Perloff D, Grim C, Flack J, et al. Human blood pressure determination by sphygmomanometry. *Circulation*. Nov 1993;88(5 Pt 1):2460-2470.
- 61. Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. *Med Care*. 1986;24:67–74.
- 62. Morisky D. E., Ang A., Krousel-Wood M, Ward, H. J. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens. 2008;10(5):348-354.
- 63. Lu, M., Safren, S. A., Skolnik, P. R., Rogers, W. H., Coady, W., Hardy, H., & Wilson, I. B. Optimal recall period and response task for self-reported HIV medication adherence. Aids and Behavior, 2008;12(1):86-94. doi:
- 10.1007/s10461-007-9261-4
- 64. Asgary R. Naderi R, Wisnivesky J. Opt-out patient navigation to improve breast and cervical cancer screening among homeless women in New York City shelters and shelter-clinics. J Womens Health (Larchmt). 2017;26(9):999-1003. doi: 10.1089/jwh.2016.6066. [Epub ahead of print].
- 65. Asgary R, Sckell B, Alcabes A, Naderi R, Ogedegbe G. Perspectives of cancer and cancer screening among homeless adults of New York City shelter-based clinics: a qualitative approach. *Cancer Causes Control*, 2015 Oct;26(10):1429-38.
- 66. Collins R, Peto R, MacMahon S, Hebert P, Fiebach NH, Eberlein KA, Godwin J, Qizilbash N, Taylor JO, Hennekens CH. Blood pressure, stroke, and coronary heart disease. Part 2, Short-term reductions in blood

pressure: overview of randomised drug trials in their epidemiological context. Lancet. 1990 Apr 7;335(8693):827-38.

- 67. Lam AY, Fresco P. Medication Adherence Measures: On Overview. Biomed Res Int. 2015; 2015:217074. doi.10.1155/2015/217074
  - 68. Voils CI, King HA, Thorpe CT, et al. Content validity and reliability of a self- report measure of medication nonadherence in hepatitis C treatment. Dig Dis Sci 2019;64:2784–97.
  - 69. Voils CI, King HA, Neelon B, et al. Characterizing weekly self- reported antihypertensive medication nonadherence across repeated occasions. Patient Prefer Adherence 2014;8:643–50.